CLINICAL TRIAL: NCT06485674
Title: Long-Term Organ Damage: Anifrolumab Versus Real-World Standard of Care in Adult Patients With Active Systemic Lupus Erythematosus (LASER) An External Comparator Arm Study for the TULIP Trials Using the University of Toronto Lupus Clinic Cohort
Brief Title: Long-Term Organ Damage: Anifrolumab Versus Real-World Standard of Care in Adult Patients With Active Systemic Lupus Erythematosus
Acronym: LASER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: D3461R00077
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Long-Term Organ Damage in Adult Patients With Active Systemic Lupus Erythematosus
Keywords: Anifrolumab; Active Systemic Lupus Erythematosus; Long-Term Organ Damage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tulip Trial Group: Patients who initiated 300 mg of anifrolumab in TULIP (Treatment of Uncontrolled Lupus via the Interferon Pathway)-1 or -2.
- Toronto Lupus Cohort Group: Participants who received RW Standard Of Care for SLE from the University of Toronto Lupus Clinic (UTLC) registry.

SUMMARY:
This is an External control arm study to generate evidence on the comparative effect of anifrolumab plus Standard of Care in TULIP versus Real World Standard of Care on organ damage in adult patients with moderately to severely active Systemic lupus erythematosus (SLE). Patients who initiated 300 mg of anifrolumab in TULIP-1 or -2 will be indexed at the date of initiating anifrolumab and will be followed up until the earliest occurrence of death, loss to follow-up, trial dis-enrollment, or week 208 assessment (in LTE study).

DETAILED DESCRIPTION:
This is an External Control arm study to generate evidence on the comparative effect of anifrolumab plus Standard of Care in TULIP versus Real World Standard of Care on organ damage in adult patients with moderately to severely active (Systemic lupus erythematosus) SLE. Patients who initiated 300 mg of anifrolumab in TULIP-1 or -2 will be indexed at the date of initiating anifrolumab and will be followed up until the earliest occurrence of death, loss to follow-up, trial dis-enrollment, or week 208 assessment (in LTE study). Patients in the University of Toronto Lupus Clinic will be indexed at the first date of clinical assessment within the patient enrollment period for which they satisfy all eligibility criteria and are receiving at least one eligible SOC treatment (i.e., their 'index assessment') and will be followed up until the earliest occurrence of death, loss to follow-up, UTLC disenrollment, or end of study period.

ELIGIBILITY:
Inclusion Criteria for UTLC:

1. Aged 18 through 70 years at index date.
2. Weight ≥40.0 kg at index date.
3. Diagnosis of paediatric or adult SLE ≥24 weeks prior to index date using ≥4 of the 11 modified ACR classification criteria at least one of which must be positive antinuclear antibody test, anti-dsDNA antibodies, or anti-Smith antibody elevated to above normal level.
4. SLEDAI-2K score ≥6 points (Table 8 in Appendix) at index date.
5. No record of current pregnancy at index date.
6. Valid measurement of SDI (Table 9 in Appendix) at index date.

Exclusion Criteria:

Selected key exclusion criteria from the TULIP trials have been adapted to the RW setting and will be applied to patients in the UTLC. Patients who meet any of the following criteria will be excluded from the study:

1. Corticosteroid dose >40 mg/day (oral prednisone equivalent) at index date.
2. Any record of receiving any biologic agent (e.g., anifrolumab, belimumab, rituximab, abatacept) at index date or within 4 weeks prior to index date.
3. Any record of malignancy at any point prior to index date, except skin malignancy ≥1 year prior to index date.
4. Record of persistent, new or recurrent nephrotic syndrome, chronic dialysis, or renal transplant at index date.
5. Serum creatinine >2.0 mg/dL (or >181 μmol/L) at index date.

   The following additional exclusion criteria may be applied to the study cohort at the time of analysis, if it is judged that their application will not significantly reduce the sample size available:
6. Record of alcohol consumption ≥14 units/week at index date or ≤1 year prior to index date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who initiated 300mg of anifrolumab in TULIP-1 or -2 will be included in the active treatment arm of this ECA study. To identify a comparator cohort of patients in the UTLC who would be considered eligible for the TULIP trials, all patients in the UTLC who were active in the database during the study time period (1 January 1995 to 31 December 2023) will be extracted,4 and all key eligibility criteria from TULIP-1 and -2 will be applied to patients in the UTLC.
Sampling Method: Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
SLICC/ACR damage index (SDI) at week 208 | 208 weeks
  Organ Damage measured using the SDI . The SDI is designed to assess irreversible damage across 12 organ systems in SLE patients, independently of cause or attribution.

SECONDARY OUTCOMES:
SDI at week 208 by organ damage at baseline | 208 weeks
  To estimate the effect of anifrolumab plus SOC in TULIP compared to RW SOC on organ damage accrual as measured by SDI at 208 weeks post-treatment initiation in the following subgroups: patients with no organ damage at baseline, and patients with any organ damage at baseline.
Time to first organ damage progression as measured by SDI. | 208 weeks
  To estimate effect of anifrolumab plus SOC in TULIP compared to RW SOC on time to first organ damage progression as measured by SDI.
Cumulative steroid intake | 208 weeks
  To estimate the effect of anifrolumab plus SOC in TULIP compared to RW SOC on cumulative steroid intake (prednisone equivalent) up to 208 weeks post-treatment initiation.
Average daily steroid dose | 208 weeks
  To estimate the effect of anifrolumab plus SOC in TULIP compared to RW SOC on average daily steroid dose (prednisone equivalent) at 208 weeks post-treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Touma, Dr, Principal Investigator — University Health Network, Toronto
Locations (1):
- Research Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No